CLINICAL TRIAL: NCT00754208
Title: Long Acting Stimulant Treatment of ADHD in Young Children
Brief Title: Long Acting Stimulant Treatment of Attention Deficit Hyperactivity Disorder (ADHD) in Young Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0380-08-FB
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Stimulant Treatment; Young Children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- methylpehnidate (Other): open-label treatment with methylphenidate
  Interventions: Drug: methylphenidate

INTERVENTIONS:
Drug: methylphenidate — Starting dose: methylphenidate (immediate-release pill) or Methylin (immediate-release chewable tablet for those unable to swallow pills) 2.5mg Q AM and Q noon. Target dose of 1mg/kg/day. Titration will occur as follows: 5mg Q AM and Q noon, then 7.5mg Q AM and Q noon, then 10mg Q AM and Q noon, as tolerated, not to exceed 30mg per day. Once each child arrives at a stable dose with a good response and good tolerability, they will be converted to the closest Ritalin LA dose, with a target dose of 1mg/kg/day.
  Other Names: Ritalin; Methylin; Ritalin LA

SUMMARY:
This is a pilot study evaluating the effectiveness, safety, and tolerability of Ritalin LA in treating Attention Deficit Hyperactivity Disorder (ADHD) in 4 and 5 year old children. Virtually no data has been published on the use of long-acting stimulant preparations in very young children despite early symptomatic development in a significant portion of young children with ADHD. This would be one of the first studies looking at a long-acting preparation of a stimulant medication in the treatment of ADHD in very young children.

Hypotheses

1. Ritalin LA is effective for the treatment of ADHD in 4 and 5 year old children.
2. Ritalin LA is reasonably well-tolerated in the treatment of ADHD in 4 and 5 year old children.

DETAILED DESCRIPTION:
This protocol involves an 8-week, open-label, pilot study evaluating the effectiveness, safety, and tolerability of Ritalin LA in treating Attention-Deficit/Hyperactivity Disorder (ADHD) in 4 and 5 year old children. The purpose of this study is to ascertain pilot data on the use of long-acting stimulants in preschool-age children since virtually no data exist on these medications in this population. The interventions include utilizing short-acting methylphenidate for the initial dosing and titration and then converting the children to Ritalin LA once an optimal dose has been found. Parents will also be receiving parent education training throughout the study. Evaluations will include obtaining the ADHD-IV at every visit, side effects of the medication, vital signs, EKG, physical exam, the Clinical Global Assessment Scale, and the Clinical Global Impression-Improvement and Severity Scales. This study will also assess parent stress with the Parent Stress Index and the emotional index of the children with the Expressed Emotion Scale for Children. Follow-up will be weekly during the first month and bi-weekly during the second month.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from the legal guardian.
* Parent and child must be English-speaking.
* The child must have been living with the parent or guardian for a minimum of 6 months at the time of study entry.
* Age: 4-5 years of age at study entry.
* weight of at least 15kg (20th percentile for 4 year olds) for boys and weight of at least 14.5kg (20th percentile for 4 year olds) for girls
* Severity: age and sex-adjusted T score greater or equal to 65 on the Hyperactive- Impulsive Subscale of both the Conners Parent and Teacher Rating Scales (L)
* Diagnosis: meets DSM-IV criteria for ADHD (hyperactive/impulsive or combined subtype), on Parent Diagnostic Interview Schedule for Children-IV (DISC-IV) and clinical interview by experienced clinician. ADHD must be the primary disorder.
* Duration: symptoms must have been present for a minimum of nine months.
* Impairment: less than or equal to 55 on the Child Global Assessment Scale.
* Cognitive functioning: An estimated IQ 70 or greater on the Peabody Picture Vocabulary Test (PPVT).
* School: participation in school-type program at least 2 half-days per week where class includes at least 8 peers; if child has been expelled from an eligible program in the 3 months before screening, they can be considered for enrollment as this may reflect severity of the disorder
* Parents and patients must be able to attend regular study visits.
* Children being treated with other stimulant or non-stimulant medications prior to enrollment will be allowed to discontinue treatment with these medications in order to enter the study, providing the parent wants to do so to enable their child to have a trial of Ritalin LA, the target symptoms are not well-controlled or unwanted side effects are persisting on their current treatment, and the prescribing physician is notified by the parent. These children will have a visit 1A in order to accommodate a 5 half-lives washout of their pre-study medication.

Exclusion Criteria:

* Other medications: no concurrent psychotropic medications or other medications (including herbal preparations and over-the-counter medications) with significant CNS effects (e.g., antidepressants, antipsychotics, drugs affecting blood pressure or heart rate, anticonvulsants, alpha-agonists, adrenergic blockers, lithium, or sedating antihistamines).
* General medical conditions: children with major medical conditions that would interfere with involvement in the study or the study medication will not be enrolled.
* Serious structural cardiac abnormalities: The recent joint advisory of the American Academy of Pediatrics (AAP) and the American Heart Association (AHA) recommend use of stimulant medications should generally be avoided in patients with cardiomyopathy, serious heart rhythm or structural abnormalities, or other serious cardiac problems. Any patient with such a diagnosis will not be allowed in this study.
* Systolic and diastolic blood pressure above 95th percentile for age and gender
* Exclusionary Psychiatric Conditions: Current Adjustment Disorder, Autism, Psychosis, Bipolar Disorder, PTSD, significant suicidality, or any other psychiatric disorder in addition to ADHD that requires treatment with additional medications.
* History of physical, sexual, or emotional abuse that results in a clinically significant impact on clinical presentation, potentially driving some of the symptoms of ADHD.
* Prior failure to respond to an adequate trial of any methylphenidate product. This will be at the determination of the investigator.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2008-09-18 (Actual); Primary Completion 2010-01-01 (Actual); Study Completion 2010-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan Daughton, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from September 2008 through Deceber 2009 in an academic medical center.
Pre-assignment Details: Please see inclusion and exclusion criteria.
Groups:
- Ritalin LA for ADHD: Subjects treated with Ritalin LA for ADHD
Period: Overall Study
Arm/Group | Ritalin LA for ADHD
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Ritalin LA for ADHD: 4 and 5 year old subjects with ADHD
Arm/Group | Ritalin LA for ADHD
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 4 [4 to 5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Child and adolescent psychiatry clinic outpatients
  Participants
    United States | 7
ADHD Subtype [Count of Participants; unit: Participants] — Diagnostic subtype identified on clinical interview and assessment of ADHD symptoms. There are a total of 18 symptoms of ADHD (9 inattentive and 9 hyperactive/impulsive). Subjects are identified as having combined subtype if >/= 6/9 inattentive and >/= 6/9 hyperactive/impulsive symptoms are endorsed. If only the inattentive criterion is met, subjects are identified as having inattentive subtype, and if only the hyperactive/impulsive criterion is met, subjects are identified as having hyperactive/impulsive subtype.
  Participants
    ADHD, combined subtype | 7
    ADHD, inattentive subtype | 0
    ADHD, hyperactive/impulsive subtype | 0
Comorbid Oppositional Defiant Disorder [Count of Participants; unit: Participants]
  YES | 4
  NO | 3
Prior Treatment [Count of Participants; unit: Participants]
  Individual therapy | 2
  Pharmacotherapy | 0
  No prior treatment | 5
Clinical Global Impression-Severity Score [Mean (Standard Deviation); unit: units on a scale] — The CGI-S is the clinician's assessment of the subject's severity of illness based upon his/her knowledge and experience with the population and disorder under study. The CGI-S is rated on a scale of 1 to 6, with 1 representing "normal, not ill", 2 representing "borderline ill", 3 representing "mildly ill", 4 representing "moderately ill", 5 representing "markedly ill", and 6 representing "severely ill."
  units on a scale | 5.14 (0.69)
Children's Global Assessment Scale [Mean (Standard Deviation); unit: units on a scale] — The children's global assessment scale is the clinician's assessment of the subject's level of functioning as rated from 0 to 100 (worst to best).
  units on a scale | 49.9 (2.04)

OUTCOME MEASURES:

1. Primary Outcome: Change in Attention Deficit Hyperactivity Disorder Rating Scale-IV Parent Version Investigator-Scored (ADHD-IV-Parent: Inv) Total Score.
Description: Change from baseline to endpoint of investigator-scored, parent version of the Attention Deficit Hyperactivity Disorder Rating Scale-IV (ADHD-IV rating scale). The ADHD-IV contains 18 items, and each item is rated 0, 1, 2 or 3. Minimum score is 0. Maximum score is 54. Change in score represents the difference between the total score at end point compared to the total score at baseline. Higher scores indicate greater symptom severity.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group 1: All subjects treated with open-label methylphenidate (Ritalin LA)
Arm/Group | Group 1
Number analyzed (Participants) | 7
units on a scale | -20.1 (13.87)

2. Secondary Outcome: Change in Clinical Global Impression-Severity
Description: Change in global rating of severity of ADHD symptoms. CGI severity is rated on a scale of 1 to 6 (normal to severely ill; refer to description in baseline information). The change in the severity rating reflects the change in this score from baseline to endpoint. The greater the reduction in score the more improvement has been observed.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group 1: All subjects treated with open-label methylphenidate
Arm/Group | Group 1
Number analyzed (Participants) | 7
units on a scale | -2.4 (1.72)

3. Secondary Outcome: Change in Children's Global Assessment Scale (CGAS) Score
Description: This measures the change in the subject's global assessment of functioning as rated by the clinician. This Children's Global Assessment Scale (CGAS) is rated on a 0-100 scale (refer to baseline information). The change in this score is the difference between the score at baseline to end point. The greater the change score, the more improvement has been observed.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1
Number analyzed (Participants) | 7
units on a scale | 9.9 (6.07)

4. Secondary Outcome: Clinical Global Impression- Improvement
Description: The Clinical Global Impression-Improvement scale is a measure of the clinician's assessment of the overall degree of improvement in ADHD symptoms from baseline to endpoint. The CGI-I is rated on a 1 to 6 scale, with 1=very much improved, 2=much improved, 3=minimally improved, 4= no change, 5= minimally worse, 6=much worse. Low numerical score on this scale indicates greater improvement.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1
Number analyzed (Participants) | 7
Participants
  Very Much Improved | 3
  Much Improved | 2
  Minimally Improved | 1
  No Change | 1
  Minimally Worse | 0
  Much Worse | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Adverse events were collected by spontaneous report
Arm/Group | Methylpehnidate
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylpehnidate (N=7)
Decreased Appetite (Gastrointestinal disorders) | 3 (3)
Irritability (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Nail biting (General disorders) | 1 (1)
Tics (Nervous system disorders) | 1 (2) — eye muscle disturbance; tongue movements

LIMITATIONS AND CAVEATS:
This study is limited by a small sample size and open-label design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No